CLINICAL TRIAL: NCT00541255
Title: Epidemiology of Asthma and Allergic Disease: Risk and Prognosis in a Cohort From Birth to Adolescence
Brief Title: A Long-Term Examination of Asthma From Childhood Through Adolescence
Status: Completed | Type: Observational
Sponsor: Isle of Wight NHS Trust (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Professor S Hasan Arshad, Chair in Allergy and Clinical Immunology, University of Southampton and Hon. Consultant Physician, University Hospital Southampton Director, The David Hide Asthma and Allergy Research Centre, Isle of Wight NHS Trust
Other Study IDs: 1408; R01HL082925 (NIH); 1R01HL082925-01A2 (NIH)
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Asthma; Dermatitis, Atopic; Rhinitis; Urticaria
Keywords: Bronchial Asthma; Food Allergy; Bronchial Hyperresponsiveness
MeSH Terms: conditions — Asthma; Dermatitis, Atopic; Rhinitis; Urticaria; Food Hypersensitivity; Bronchial Hyperreactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, saliva, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Asthma is a common disease that is often diagnosed in childhood. In some teenagers, asthma symptoms disappear and treatment can be stopped; however, for some of these people, asthma symptoms return in adulthood. This study will examine data collected over the lifetime of 18-year olds to identify factors that may increase a person's chance of having recurrent asthma as an adult.

DETAILED DESCRIPTION:
Asthma is a serious, long-term illness that affects around 15% of children in the United States. During adolescence, up to 50% of teenagers stop experiencing symptoms and are able to discontinue treatment. However, asthma symptoms often reoccur in adulthood for many of these people. It is not known exactly what causes this recurrence, but potential risk factors may include obesity, elevated serum leptin levels, early onset of puberty, exposure to pollutants, parental smoking habits, and lack of breastfeeding. Additionally, it is not known why childhood asthma is initially more prevalent in boys, but during adolescence it becomes more prevalent in girls. Beginning in 1989, a group of children born on the Isle of Wight in the United Kingdom has been followed by study researchers to provide long-term information on asthma. These children have been periodically evaluated over the years and are now 18 years old. The purpose of this study is to analyze participants' data collected over a span of 18 years to identify factors that may increase a person's risk of experiencing persistent or recurrent asthma in adulthood.

At previous study visits that occurred when participants were 1, 2, 4, and 10 years old, information on the following was collected: asthma and other allergic diseases, family history of asthma, and early life risk factors, including breastfeeding and tobacco smoke exposure. A blood sample was collected at participants' 10-year study visit. For this current study, all 18-year-old participants will return for a study visit. Participants will complete questionnaires on asthma and allergy symptoms and environmental exposures, including tobacco smoke and pollution. Blood collection, an allergy skin prick test, lung function testing, and a bronchial challenge test to assess airway function will occur. Select participants will also have a sputum sample collected.

ELIGIBILITY:
Inclusion Criteria:

* Born on the Isle of Wight in the United Kingdom between January 1, 1989 and February 28, 1990

Exclusion criteria:

* Refused consent

Ages: 17 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consists of around 1500 unselected subjects (now age 18) who were recruited at birth. This is a homogenous population with 99% being Caucasians.
Sampling Method: Non-Probability Sample
Enrollment: 1313 (Actual)
Dates: Start 2007-09; Primary Completion 2012-05 (Actual); Study Completion 2015-02-18 (Actual)

PRIMARY OUTCOMES:
Identifying factors that may increase a person's chance of having recurrent asthma as an adult | Measured throughout the participant's lifetime

CONTACTS AND LOCATIONS:
Overall Officials: Syed Arshad, MD, Principal Investigator — University of Southampton, United Kingdom
Locations (1):
- The David Hide Asthma and Allergy Research Centre, Newport, Isle Of Wight, United Kingdom

REFERENCES:
- See also: Click here for The David Hide Asthma and Allergy Research Centre Web site — http://www.davidhideallergyresearch.co.uk